CLINICAL TRIAL: NCT00287534
Title: A Prospective, Multi-Centre, Randomised, Open Parallel Group Study to Compare the Effectiveness and Compatibility of ARIMIDEX (ZD 1033) With NOLVADEX After a Prior 2 Years' Treatment With Tamoxifen in Adjuvant Therapy of Breast Carcinoma in Postmenopausal Women.
Brief Title: Effectiveness of Combination of Arimidex and Nolvadex in Adjuvant Therapy of Breast Carcinoma in Postmenopausal Women.
Acronym: ARNO-95
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: German Adjuvant Breast Cancer Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1033GR/0001; ARNO-95
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

ARMS (2):
- 1 (Experimental): Anastrozole
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Tamoxifen
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — oral
  Other Names: Arimidex; ZD1033
  Arms: 1
Drug: Tamoxifen — oral
  Other Names: Nolvadex
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy and tolerability of 3 years treatment with anastrozole after a prior 2 years' treatment with tamoxifen versus 5 years treatment with tamoxifen in postmenopausal women with early breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Post-menopausal women ≤75 years,
* histologically confirmed invasive breast carcinoma (no distant metastases),
* positive hormone receptor status,
* continuous 2-year adjuvant tamoxifen therapy 20 mg/30 mg with 4 weeks after primary surgery

Exclusion Criteria:

* menopause status maintained by medication,
* pre-operative chemotherapy or hormone therapy or radiation therapy,
* relapse or second carcinoma or previous cancerous disease,
* breast carcinoma in situ,
* simultaneous carcinoma of the opposite side or secondary breast,
* 10 or more tumour-infiltrated lymph nodes.
* serious accompanying diseases

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1059 (Estimated)
Dates: Start 1996-11; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To assess the difference in disease-free survival between post-menopausal women with hormone receptor-positive early breast cancer who switched from tamoxifen to anastrozole and those who continued to receive tamoxifen

SECONDARY OUTCOMES:
To assess difference in overall survival between the two treatment arms
To assess difference in disease recurrence between the two treatment arms
To assess difference in safety and tolerability between the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Kaufmann, MD, Principal Investigator — German Adjuvant Breast Cancer Group
Locations (43):
- Germany (43):
  - Research Site, Albstadt
  - Research Site, Berlin
  - Research Site, Cloppenburg
  - Research Site, Eggenfelden
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanau
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Hoyerswerda
  - Research Site, Idar-Oberstein
  - Research Site, Jena
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Leonberg
  - Research Site, Lingen
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Münster
  - Research Site, Neustadt
  - Research Site, Osnabrück
  - Research Site, Paderborn
  - Research Site, Pforzheim
  - Research Site, Recklinghausen
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Rüsselsheim am Main
  - Research Site, Schleswig
  - Research Site, Siegen
  - Research Site, Titisee-Neustadt
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Waiblingen
  - Research Site, Westerstede
  - Research Site, Worms
  - Research Site, Würzburg